CLINICAL TRIAL: NCT01688739
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 334 in Healthy Subjects and Migraine Patients
Brief Title: Ascending Single Doses of Erenumab (AMG 334) in Healthy Adults and Migraine Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20101267; 2011-005600-15 (EudraCT Number)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erenumab (Experimental): Participants received a single dose of erenumab by subcutaneous injection at doses of 1 mg, 7 mg, 21 mg, 70 mg, 140 mg, and 210 mg or by IV injection at a dose of 140 mg.
  Interventions: Drug: Erenumab
- Placebo (Placebo Comparator): Participants received a single dose of matching placebo administered by SC or IV injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erenumab — Administered by subcutaneous injection or intravenous injection
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab
Drug: Placebo — Administered by subcutaneous injection or intravenous injection
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether erenumab is safe and well tolerated in healthy adults and migraine patients. As part of the secondary objectives, this study will be conducted to characterize the pharmacokinetic (PK) profile of erenumab after single subcutaneous (SC) or intravenous (IV) doses in healthy participants and migraine patients as well as to characterize the effect of erenumab on the capsaicin-induced increase in dermal blood flow after single SC or IV doses in healthy participants and migraine patients.

DETAILED DESCRIPTION:
This study was a single-dose, double-blind, placebo-controlled, sequential dose escalation study in which participants were to be enrolled into 8 cohorts.

In Part 1 healthy participants were randomized in a 3:1 ratio (erenumab:placebo) into 6 cohorts: 5 cohorts received the investigational product (IP) as an SC administration and 1 cohort received it as an IV administration. In Part 2 a total of 12 migraine patients were randomized in a 1:1 ratio (erenumab:placebo) in cohort 7. An additional 8 migraine patients could have been enrolled and randomized in a 3:1 ratio in the optional cohort 8, however this cohort was not enrolled.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female subjects between 18 and 45 years of age, or male or female subjects with migraines between 18 and 55 years of age, inclusive, with no history or evidence of clinically relevant medical disorders as determined by the investigator in consultation with the Amgen physician;

Exclusion Criteria:

- History or evidence of clinically significant disorder (including psychiatric), condition or disease that, in the opinion of the Investigator or Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2013-03-27 (Actual); Study Completion 2013-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Leuven, Belgium

REFERENCES:
- [Background] Vu T, Ma P, Chen JS, de Hoon J, Van Hecken A, Yan L, Wu LS, Hamilton L, Vargas G. Pharmacokinetic-Pharmacodynamic Relationship of Erenumab (AMG 334) and Capsaicin-Induced Dermal Blood Flow in Healthy and Migraine Subjects. Pharm Res. 2017 Sep;34(9):1784-1795. doi: 10.1007/s11095-017-2183-6. Epub 2017 Jun 7. PMID 28593473
- [Background] de Hoon J, Van Hecken A, Vandermeulen C, Yan L, Smith B, Chen JS, Bautista E, Hamilton L, Waksman J, Vu T, Vargas G. Phase I, Randomized, Double-blind, Placebo-controlled, Single-dose, and Multiple-dose Studies of Erenumab in Healthy Subjects and Patients With Migraine. Clin Pharmacol Ther. 2018 May;103(5):815-825. doi: 10.1002/cpt.799. Epub 2017 Oct 24. PMID 28736918
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Belgium from March 2012 to March 2013.
  The study enrolled healthy participants (Part 1) and participants who had migraines for at least 6 months and at least 3 migraine attacks per month in the last 3 months (Part 2).
Pre-assignment Details: Healthy participants were randomized in a 3:1 ratio to erenumab or placebo within each dose cohort. Migraine participants were randomized in a 1:1 ratio to erenumab or placebo.
Groups:
- Healthy: Placebo: Healthy participants received a single dose of matching placebo administered by subcutaneous (SC) or intravenous (IV) injection.
- Healthy: Erenumab 1 mg SC: Healthy participants received a single dose of erenumab 1 mg administered by subcutaneous injection.
- Healthy: Erenumab 7 mg SC: Healthy participants received a single dose of erenumab 7 mg administered by subcutaneous injection.
- Healthy: Erenumab 21 mg SC: Healthy participants received a single dose of erenumab 21 mg administered by subcutaneous injection.
- Healthy: Erenumab 70 mg SC: Healthy participants received a single dose of erenumab 70 mg administered by subcutaneous injection.
- Healthy: Erenumab 140 mg SC: Healthy participants received a single dose of erenumab 140 mg administered by subcutaneous injection.
- Healthy: Erenumab 140 mg IV: Healthy participants received a single dose of erenumab 140 mg administered by intravenous injection.
- Healthy: Erenumab 210 mg SC: Healthy participants received a single dose of erenumab 210 mg administered by subcutaneous injection.
- Migraine: Placebo: Participants with migraine received a single dose of placebo administered by subcutaneous injection.
- Migraine: Erenumab 140 mg SC: Participants with migraine received a single dose of erenumab 140 mg administered by subcutaneous injection.
Period: Overall Study
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC
Started | 13 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Received Study Drug | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC | Total
Number analyzed (Participants) | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for each part of the study.
  years
    Healthy Participants: number analyzed (Participants) | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 48
    Healthy Participants | 28.6 (6.1) | 22.0 (1.7) | 26.0 (7.9) | 25.7 (6.9) | 27.5 (6.6) | 28.0 (8.5) | 31.0 (8.1) | 26.2 (7.0) |  |  | 27.4 (6.8)
    Migraine Participants: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 12
    Migraine Participants |  |  |  |  |  |  |  |  | 28.5 (12.6) | 23.8 (5.4) | 26.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 9
  Male | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 1 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 12 | 3 | 3 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 3 | 3 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment. The definition of adverse events includes worsening of a pre-existing medical condition. Laboratory value changes that require treatment or adjustment in current therapy are considered adverse events.
  Teatment-related adverse events (TRAEs) are those assessed by the investigator as being possibly related to study drug.
  A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal
  * life-threatening (places the subject at immediate risk of death)
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From the initial dose of study drug up to 155 days.
Population: All participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Any adverse event | 10 | 2 | 1 | 6 | 5 | 5 | 5 | 6 | 5 | 6
  Serious adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 4 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies
Description: Participants who had a negative or no result at baseline and were antibody positive postbaseline. Blood samples were first tested for anti-erenumab binding antibodies, samples testing positive for binding antibodies were also tested for neutralizing antibodies.
Time Frame: Baseline and up to 155 days postdose
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Binding antibody positive | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutralizing antibody positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Erenumab
Time Frame: Predose to 155 days postdose
Population: All participants who received erenumab
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL | 0.0077 (0.00395) | 0.302 (0.145) | 1.17 (0.646) | 6.25 (2.03) | 9.18 (1.97) | 47.8 (4.09) | 15.2 (4.78) | 9.93 (3.42)
Statistical Analysis 1: Comparison: Healthy: Erenumab 140 mg SC vs Migraine: Erenumab 140 mg SC; Test type: Other; p = 0.7595, ANCOVA; Ratio of Geometric Means = 1.1, 90% CI 2-sided [0.8 to 1.4] — Migraine participants / Healthy Participants

4. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Erenumab
Time Frame: Predose to 155 days postdose
Population: All participants who received erenumab
Measure: Median (Full Range); unit: days
Arm/Group | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6
days | 4.0 [2.0 to 7.0] | 7.0 [4.0 to 7.0] | 7.0 [3.0 to 10] | 6.0 [3.0 to 11] | 5.5 [4.0 to 21] | 0.069 [0.069 to 0.38] | 8.5 [4.0 to 11] | 11 [7.0 to 14]

5. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Erenumab
Time Frame: Predose to 155 days postdose
Population: All participants who received erenumab
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6
days*µg/mL | 0.0851 (0.0169) | 4.01 (2.07) | 23.5 (15.5) | 171 (60.9) | 332 (57.9) | 614 (112) | 652 (221) | 367 (102)
Statistical Analysis 1: Comparison: Healthy: Erenumab 140 mg SC vs Migraine: Erenumab 140 mg SC; Test type: Other; p = 0.5481, ANCOVA; Ratio of Geometric Means = 1.1, 90% CI 2-sided [0.9 to 1.4] — Migraine participants / Healthy participants

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of Erenumab
Time Frame: Predose to 155 days postdose
Population: All participants who received erenumab
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 0 | 3 | 6 | 6 | 6 | 6 | 6 | 6
days*µg/mL |  | 4.13 (2.04) | 24.5 (17.0) | 174 (78.6) | 333 (57.9) | 615 (112) | 653 (222) | 367 (103)
Statistical Analysis 1: Comparison: Healthy: Erenumab 140 mg SC vs Migraine: Erenumab 140 mg SC; Test type: Other; p = 0.5506, ANCOVA; Ratio of Geometric Means = 1.1, 90% CI 2-sided [0.9 to 1.4] — Migraine participants / Healthy participants

7. Secondary Outcome: Ratio of Post-capsaicin Dermal Blood Flow to Pre-capsaicin Dermal Blood Flow
Description: Inhibition of capsaicin-induced dermal blood flow (DBF) by erenumab was used to measure calcitonin gene-related peptide (CGRP) receptor antagonism. Capsaicin was applied at 2 sites on the volar surface of the participants' left or right forearms and a control mixture was applied to 1 site on the volar surface of either the participants' left or right forearm. Dermal blood flow was assessed by laser Doppler perfusion imaging and was done immediately before ('baseline') and 0.5 hours post-capsaicin on the surface of these 3 sites.
  Data reported are the least square geometric mean ratios for the post-capsaicin dermal blood flow to pre-capsaicin dermal blood flow.
  According to the protocol, not all cohorts had dermal blood flow measurements at all time points.
Time Frame: Days 4, 15, 29, 43, 64, 85, 99, 127, and end of study (defined as day 43 for the 1 mg, 7 mg and 21 mg erenumab cohorts, day 99 for the 70 mg erenumab cohort, day 127 for the 140 mg erenumab cohorts and day 155 for the 210 mg erenumab cohort).
Population: All participants for whom at least one post-dose capsaicin response measure was recorded.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC
Number analyzed (Participants) | 12 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ratio
  Day 4 | 8.6 (1.15) | 9.9 (1.32) | 5.6 (1.32) | 2.9 (1.22) | 1.7 (1.22) | 1.4 (1.22) | 1.4 (1.22) | 1.9 (1.22) | 11.9 (1.20) | 2.0 (1.20)
  Day 15 | 8.6 (1.15) | 9.0 (1.32) | 3.6 (1.32) | 1.4 (1.22) | 2.2 (1.22) | 1.3 (1.22) | 1.7 (1.22) | 2.2 (1.22) | 12.4 (1.20) | 2.1 (1.20)
  Day 29 | 7.2 (1.15) | 8.3 (1.32) | 10.8 (1.32) | 3.0 (1.22) | 2.0 (1.22) | 1.1 (1.22) | 1.6 (1.22) | 1.9 (1.22) | 13.1 (1.20) | 1.8 (1.20)
  Day 43: number analyzed (Participants) | 12 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
  Day 43 | 8.4 (1.19) |  |  |  | 1.2 (1.26) | 1.8 (1.22) | 2.0 (1.22) | 2.1 (1.22) | 12.0 (1.20) | 2.1 (1.20)
  Day 64: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Day 64 | 8.3 (1.21) |  |  |  |  | 1.5 (1.22) | 2.2 (1.22) | 2.3 (1.22) | 12.4 (1.20) | 2.0 (1.20)
  Day 85: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Day 85 | 10.7 (1.21) |  |  |  |  | 4.6 (1.26) | 3.9 (1.22) | 2.6 (1.22) | 12.0 (1.20) | 7.4 (1.20)
  Day 99: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Day 99 | 7.6 (1.21) |  |  |  |  | 5.1 (1.22) | 5.9 (1.22) | 4.3 (1.22) | 12.2 (1.20) | 10.2 (1.20)
  Day 127: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
  Day 127 | 11.4 (1.36) |  |  |  |  |  |  | 9.1 (1.22) |  |
  End of study | 9.6 (1.15) | 8.2 (1.32) | 10.5 (1.32) | 9.0 (1.22) | 3.6 (1.22) | 7.6 (1.22) | 8.3 (1.22) | 8.8 (1.22) | 12.0 (1.20) | 9.8 (1.20)

ADVERSE EVENTS:
Time Frame: From the initial dose of study drug up to 155 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Healthy: Placebo | Healthy: Erenumab 1 mg SC | Healthy: Erenumab 7 mg SC | Healthy: Erenumab 21 mg SC | Healthy: Erenumab 70 mg SC | Healthy: Erenumab 140 mg SC | Healthy: Erenumab 140 mg IV | Healthy: Erenumab 210 mg SC | Migraine: Placebo | Migraine: Erenumab 140 mg SC
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 10/12 | 2/3 | 1/3 | 6/6 | 5/6 | 5/6 | 5/6 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy: Placebo (N=12) | Healthy: Erenumab 1 mg SC (N=3) | Healthy: Erenumab 7 mg SC (N=3) | Healthy: Erenumab 21 mg SC (N=6) | Healthy: Erenumab 70 mg SC (N=6) | Healthy: Erenumab 140 mg SC (N=6) | Healthy: Erenumab 140 mg IV (N=6) | Healthy: Erenumab 210 mg SC (N=6) | Migraine: Placebo (N=6) | Migraine: Erenumab 140 mg SC (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 3
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 1 | 1 | 2 | 4 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.